CLINICAL TRIAL: NCT01177618
Title: Genetic Epidemiology of Severe, Early-Onset Chronic Obstructive Pulmonary Disease
Brief Title: Boston Early-Onset Chronic Obstructive Pulmonary Disease (COPD) Study
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Edwin K. Silverman, Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 1437; U01HL089856 (NIH); NCT00106444 (obsolete NCT alias)
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Emphysema; Chronic Bronchitis; Genetics; Association Studies
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA, Serum, Plasma, Buccal Brushings, and Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Probands: Severe, early-onset COPD subjects that bring the family into the study
- Relatives: Relatives of early-onset COPD probands, including first-degree relatives (parents, siblings, and children), second-degree relatives (aunts, uncles, grandparents, half-siblings), spouses, and other affected individuals.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is often caused by cigarette smoking, but genetic predisposition also influences COPD susceptibility. The purpose of this study is to identify genetic factors that predispose some individuals to develop COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD), which is the third leading cause of death in the United States, affects millions of people around the world. COPD, which can include both emphysema and chronic bronchitis, affects the lungs making it very difficult to breathe. Cigarette smoking is the most common risk factor for developing COPD; however, only 15% to 20% of smokers develop COPD in their lifetimes. The onset of COPD also varies greatly from person to person; while some people do not develop respiratory symptoms until later in life, there are others who develop severe COPD at a very early age. Prior research has led to the discovery of the alpha-1 antitrypsin protein deficiency in association with COPD development. This discovery has generated further interest toward studying other genetic factors which may also affect an individual's likelihood of developing COPD. Therefore, the purpose of the Boston Early-Onset COPD study is to gain a better understanding of COPD risk factors in order to establish new possible methods of treatment for people affected by COPD.

For this study we are enrolling individuals affected with severe COPD (52 years old or younger with an FEV1 < 40%) and their family members. Each participant will attend one study visit that involves a respiratory questionnaire, a breathing test, and blood draw. This visit can be completed at the participant's home, in the hospital, or by long distance data collection (phone interview, local breathing tests, and local blood draw with mailed samples), whichever is preferred.

ELIGIBILITY:
Inclusion Criteria for Early-Onset COPD Probands:

* Early onset of COPD in individuals younger than 53 years old
* Spirometry results that are indicative of severe COPD (FEV1 < 40% predicted)
* Physician-diagnosed COPD

Exclusion Criteria for Early-Onset COPD Probands:

* Severe alpha-1 antitrypsin deficiency
* Other chronic lung diseases in participants with COPD (except asthma)
* Pregnant
* Any previous lung surgery including lung transplant or lung reduction volume surgery (LVRS); unless prior Pulmonary Function Tests are available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Severe, early-onset COPD subjects and their relatives
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 1994-07; Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
No Primary Outcome | Single Visit for approximately two hours to collect study data and samples
  Since this is an observational study, there are no primary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Edwin K. Silverman, M.D., Ph.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
For subjects approved for data sharing by our IRB, we will release genome sequencing data through dbGaP.
Supporting Information: Analytic Code
Time Frame: dbGaP submission is being performed by TOPMed for eligible subjects. Although TOPMed controls this data release, it typically occurs within six months of data generation.
Access Criteria: Approval through dbGaP

REFERENCES:
- [Result] Cho MH, Ciulla DM, Klanderman BJ, Hersh CP, Litonjua AA, Sparrow D, Raby BA, Silverman EK. Analysis of exonic elastin variants in severe, early-onset chronic obstructive pulmonary disease. Am J Respir Cell Mol Biol. 2009 Jun;40(6):751-5. doi: 10.1165/rcmb.2008-0340OC. Epub 2008 Nov 21. PMID 19029017
- [Result] Hersh CP, DeMeo DL, Al-Ansari E, Carey VJ, Reilly JJ, Ginns LC, Silverman EK. Predictors of survival in severe, early onset COPD. Chest. 2004 Nov;126(5):1443-51. doi: 10.1378/chest.126.5.1443. PMID 15539711
- [Result] DeMeo DL, Reilly JJ, Ginns LC, Sylvia JS, Silverman EK. Concordance of genotypes in pre- and post-lung transplantation DNA samples. Am J Respir Cell Mol Biol. 2005 Oct;33(4):402-5. doi: 10.1165/rcmb.2005-0142OC. Epub 2005 Jun 30. PMID 15994430
- [Result] DeMeo DL, Carey VJ, Chapman HA, Reilly JJ, Ginns LC, Speizer FE, Weiss ST, Silverman EK. Familial aggregation of FEF(25-75) and FEF(25-75)/FVC in families with severe, early onset COPD. Thorax. 2004 May;59(5):396-400. doi: 10.1136/thx.2003.012856. PMID 15115866
- [Result] Silverman EK, Palmer LJ, Mosley JD, Barth M, Senter JM, Brown A, Drazen JM, Kwiatkowski DJ, Chapman HA, Campbell EJ, Province MA, Rao DC, Reilly JJ, Ginns LC, Speizer FE, Weiss ST. Genomewide linkage analysis of quantitative spirometric phenotypes in severe early-onset chronic obstructive pulmonary disease. Am J Hum Genet. 2002 May;70(5):1229-39. doi: 10.1086/340316. Epub 2002 Mar 25. PMID 11914989
- [Result] Silverman EK, Weiss ST, Drazen JM, Chapman HA, Carey V, Campbell EJ, Denish P, Silverman RA, Celedon JC, Reilly JJ, Ginns LC, Speizer FE. Gender-related differences in severe, early-onset chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2000 Dec;162(6):2152-8. doi: 10.1164/ajrccm.162.6.2003112. PMID 11112130
- [Result] Silverman EK, Chapman HA, Drazen JM, Weiss ST, Rosner B, Campbell EJ, O'DONNELL WJ, Reilly JJ, Ginns L, Mentzer S, Wain J, Speizer FE. Genetic epidemiology of severe, early-onset chronic obstructive pulmonary disease. Risk to relatives for airflow obstruction and chronic bronchitis. Am J Respir Crit Care Med. 1998 Jun;157(6 Pt 1):1770-8. doi: 10.1164/ajrccm.157.6.9706014. PMID 9620904